CLINICAL TRIAL: NCT04714294
Title: To Evaluate the Safety, Tolerability, Pharmacokinetics Characteristics of HPP737 in Healthy Volunteers: a Randomized, Double-blind, Placebo-controlled, Dose Escalation Phase I Clinical Study
Brief Title: Evaluate the Safety, Tolerability and Pharmacokinetics Characteristics of HPP737 in Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Newsoara Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Newsoara HYK Biopharmaceutical (Shanghai) Co., Ltd. (Industry)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HPP737-PK-103
Record Dates: First submitted 2020-12-18; First posted 2021-01-19 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2020-12

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: SAD: planned 48 arms. 12 subjects each arm (Active: placebo=3:1) MAD: planned 36 arms. 12 subjects each arm (Active: placebo=3:1)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SAD: Each volunteer will receive 6 mg, 10mg, 20mg, 40mg(or TBD) of IP once daily for 1 day (Experimental): Drug: HPP737 or placebo One 1 mg capsule and one 5mg capsule taken orally (by mouth) once daily for SAD arm 1/ Two 5mg capsule taken orally (by mouth) once daily for SAD arm 2/ Four 5mg capsule taken orally (by mouth) once daily for SAD arm 3/ Eight 5mg capsule taken orally (by mouth) once daily for SAD arm 4
  Interventions: Drug: HPP737 or placebo
- MAD: Each volunteer will receive 10mg, 20mg, 40mg(or TBD) of IP once daily for 7 days (Experimental): Drug: HPP737 or placebo Two 5mg capsule taken orally (by mouth) once daily for MAD arm 1/ Four 5mg capsule taken orally (by mouth) once daily for MAD arm 2/ Eight 5mg capsule taken orally (by mouth) once daily for MAD arm 3
  Interventions: Drug: HPP737 or placebo

INTERVENTIONS:
Drug: HPP737 or placebo — HPP737 or placebo will be randomized to assign to subjects

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a common, preventable and treatable disease characterized by persistent respiratory symptoms and incompletely reversible airflow limitation. It is usually caused by airway and / or alveolar abnormalities caused by obvious exposure to toxic particles or gases.COPD is currently the fourth leading cause of death in the world, and is expected to be the third leading cause of death by 2020.HPP737 as an oral PDE4 inhibitor for the treatment of COPD.Preclinical data showed that the activity of HPP737 was similar to that of rofloxacin, but HPP737 significantly reduced the permeability to CNS and may have better tolerance. HPP737 will be used to develop indications for chronic obstructive pulmonary disease, and PK study in Chinese people is going to to evaluate the safety and tolerability of HPP737 in healthy volunteers.

DETAILED DESCRIPTION:
This PK study it to evaluate the safety and tolerability of HPP737 in healthy subjects.

84 healthy subjects were included.A single dose of about 48 patients: expected 6mg, 10mg, 20mg, 40mg or undetermined, 12 subjects in each group, the ratio of HPP737 to placebo was 3:1 (9 cases: 3 cases), 6mg and 10mg could be carried out simultaneously.The dose group and the total number of subjects can be adjusted according to the latest data obtained.

There were 36 patients with multiple doses: expected 10mg, 20mg, 40mg or undetermined, with 12 subjects in each group. The ratio of HPP737 to placebo was 3:1 (9 cases: 3 cases). The dose group and total number of subjects could be adjusted according to the latest data. Multiple dose group and single dose group can be carried out simultaneously. Each multiple dose group will be enrolled after the first subject in the same dose group of single dose is enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent and participated in the study voluntarily;
2. Male and female aged 45 to 18 years old;
3. Male or female who agree to take effective contraception from the screening period to 90 days after the last medication of the trial, and agree to take at least one effective contraceptive measure;
4. In the screening and baseline period, the body weight of male was no less than 50kg, and that of female was no less than 45kg. Body mass index (BMI) was in the range of 19-24kgm2(including 19 and 24), [BMI = weight (kg)) height2(M2)];

Exclusion Criteria:

1. Have specific allergic history or allergic constitution such as drugs, food, pollen, etc., or be allergic to PDE4 inhibitors or similar drugs;
2. Patients with previous diseases of neuropsychiatric system, respiratory system, cardiovascular system, digestive system, haemolymph system, liver and kidney system, endocrine system, skeletal muscle system or other diseases, and the investigator judged that the previous medical history may have an impact on drug metabolism or safety;
3. Screening or baseline showing abnormal vital signs, physical examination, laboratory examination, electrocardiogram and other results with clinical significance;
4. Patients with history of malignant tumor in the past 5 years;
5. Abnormal chest X-ray or abdominal B-ultrasound with clinical significance;
6. Patients with positive HBsAg, HCV antibody, HIV antibody or syphilis antibody;
7. Having a history of drug dependence or drug abuse, or positive urine drug abuse screening;
8. Smokers (5 or more cigarettes a day);
9. Alcoholics (drinking more than 14 units per week, each unit is equivalent to 360ml beer or 150ml wine or 45ml liquor with 40% alcohol volume);

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2020-09-08 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate changes of Safety and tolerability from day 1 to day 7 (SAD) or day 14(MAD) | SAD: from the screening period to the 7th day; MAD: from the screening period to the 14th day;
  Incidence and severity of various adverse events, including physical examination, blood routine, blood biochemistry, urine flow sediment test, coagulation function, vital signs (pulse, respiration, blood pressure, body temperature), electrocardiogram, etc

SECONDARY OUTCOMES:
Evaluate changes of Pharmacokinetics (PK) evaluation mainly Cmax from day 1 to day 7 (SAD) or day 14 (MAD) | SAD: from the screening period to the 7th day; MAD: from the screening period to the 14th day;
  Plasma HPP737 concentration and pharmacokinetic parameters：Cmax

OTHER OUTCOMES:
Evaluate changes of Pharmacokinetics (PK) evaluation mainly AUC0-24 from day 1 to day 7 (SAD) or day 14 (MAD) | SAD: from the screening period to the 7th day; MAD: from the screening period to the 14th day;
  Plasma HPP737 concentration and pharmacokinetic parameters： AUC0-24

CONTACTS AND LOCATIONS:
Overall Officials: Nengming Lin, Dr, Principal Investigator — Hangzhou, Zhejiang Province
Locations (1):
- Affiliated Hangzhou First People's Hospital.Zhejiang University School of Medicine, Hangzhou, Zhejiang, China